CLINICAL TRIAL: NCT00268593
Title: A Randomised Phase II Study of Two Dose Schedules of PI-88 in Combination With Docetaxel in Patients With Androgen-independent Prostate Cancer
Brief Title: Pilot Efficacy Study of PI-88 With Docetaxel to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Progen Pharmaceuticals (Industry)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other); Aventis Pharmaceuticals (Industry)
Responsible Party: Darryn Bampton, Progen Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR88206; PROPIT; XRP6976J/6216
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
Keywords: heparanase; angiogenesis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — phosphomannopentaose sulfate; Docetaxel; Prednisone

ARMS (2):
- 130 mg PI-88 + docetaxel (Experimental): 130 mg PI-88 7 days/week + docetaxel 75 mg/m2
  Interventions: Drug: PI-88; Drug: docetaxel; Drug: prednisone
- 250 mg PI-88 + docetaxel (Experimental): 250 mg PI-88 4 days/week + docetaxel 75 mg/m2
  Interventions: Drug: PI-88; Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: PI-88 — Subcutaneous injection administered 7 days/week for 130 mg PI-88 and 4 days/week for 250 mg PI-88; patients to be treated until progression or withdrawal from study.
Drug: docetaxel — Subcutaneous injection administered 7 days/week for 130 mg PI-88 and 4 days/week for 250 mg PI-88; patients to be treated until progression or withdrawal from study.
Drug: prednisone — 5 mg twice a day orally

SUMMARY:
Docetaxel (Taxotere) is an approved chemotherapeutic drug for the treatment of androgen-independent prostate cancer. The aim of the study is to investigate whether addition of the investigational drug PI-88 will increase the efficacy of docetaxel in this disease. PI-88 inhibits cancer growth by inhibiting the development of new blood vessels and starving the tumour of oxygen and nutrients (anti-angiogenic). Because PI-88 and docetaxel have different mechanisms of action, they are expected to have increased (synergistic) activity when combined.

DETAILED DESCRIPTION:
The trial is a multi-centre, open-label randomised phase II study in patients with androgen-independent prostate cancer (AIPC), with a lead-in combination tolerance study. The aim of the lead-in phase is to establish the maximum tolerated dose (MTD) of PI-88 administered either 4 days/week or 7 days/week) in combination with fixed doses of docetaxel (75 mg/m^2 every 21 days) and prednisone (5 mg twice daily). In the randomized phase II component, patients will receive PI-88 at the MTD, either 4 days/week or 7 days/week, in combination with docetaxel and prednisone. The patients will receive up to 10 treatment cycles of the combination therapy. Response to treatment will be assessed by measuring serum levels of prostate specific antigen (PSA). Other efficacy measures will include radiological assessment, progression-free survival, overall survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven prostate adenocarcinoma that is unresponsive or refractory to hormone therapy
* Patients must have received prior hormonal therapy, defined as castration by orchiectomy and/or luteinizing hormone releasing hormone (LHRH) agonists
* Patients must have documented progression detected by PSA increase, physical examination and/or imaging
* Patients must have achieved stable pain control for a minimum of seven consecutive days prior to study entry.
* Prior radiation therapy (to < 25% of the bone marrow only) is permitted. At least 4 weeks must have elapsed since the completion of radiation therapy and the patient must have recovered from side effects prior to study entry.
* Prior surgery is allowed. At least 4 weeks must have elapsed since the completion of surgery
* Life expectancy > 3 months
* ECOG Performance score of < 2.
* Neutrophil count > 1.5 x 109/L (1,500/mm3)
* Haemoglobin > 10 g/dL
* Platelet count > 100 x 109/L (100,000/mm3)
* Total bilirubin < the upper limit of normal (ULN) of the institution
* ALT (SGPT) and AST (SGOT) < 1.5 x the ULN of the institution
* Calculated creatinine clearance, using Cockroft and Gault formula, >60 mL/min
* APTT and PT < 1.5 X ULN
* Patients (or legally acceptable representative) must have voluntarily given written informed consent to participate in this study.
* Patients must be willing to comply with the scheduled visit, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Prior cytotoxic chemotherapy
* Prior isotope therapy (e.g., strontium, samarium)
* Prior radiotherapy to >25% of bone marrow (whole pelvic irradiation is not allowed)
* Prior treatment with biological response modifiers within the previous 4 weeks
* Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, or any other cancer from which the patient has been disease-free for > 5 years
* Known brain or leptomeningeal involvement
* Symptomatic peripheral neuropathy > grade 2 according to the NCI Common Terminology Criteria for Adverse Events v3 (NCI CTCAE v3)
* Serious intercurrent medical illness that does not permit adequate follow-up and compliance with the study protocol
* History of immune-mediated thrombocytopenia, thrombotic thrombocytopenic purpura or other platelet disease, or laboratory evidence of anti-heparin antibodies
* Use of drugs that may inhibit the metabolism of docetaxel (cyclosporin, terfenadine, ketoconazole, erythromycin, troleandomycin) within the previous week or during the study
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study screening
* Treatment with any other anti-cancer therapy (except LHRH agonists) including any prescribed compounds and/or over-the-counter (OTC) products for the treatment of prostate cancer must be stopped prior to day of enrolment
* Treatment with systemic corticosteroids used for reasons other than specified by the protocol must be stopped prior to day of enrolment
* Concomitant bisphosphonate therapy is not allowed. Patients already receiving bisphosphonates must be stopped prior to day of enrolment
* Concomitant use of aspirin (> 150 mg/day), non-steroidal anti-inflammatory drugs (except specific COX-2 inhibitors), heparin, low molecular weight heparin (LMWH), warfarin (> 1 mg/day) or anti-platelet drugs (abciximab, clopidogrel, dipyridamole, ticlopidine and tirofiban). Low-dose aspirin (≤ 150 mg/day) and low-dose warfarin (≤ 1 mg/day) are permitted as concomitant medications
* Treatment with heparin or low molecular weight heparin within the previous two weeks is not permitted
* History of allergy and/or hypersensitivity to heparin or other anti-coagulants/thrombolytic agents
* History of acute or chronic gastrointestinal bleeding within the last two years, inflammatory bowel disease or other abnormal bleeding tendency
* Patients at risk of bleeding due to open wounds or planned surgery
* Myocardial infarction, stroke or congestive heart failure within the past three months
* Uncontrolled or serious infection within the past four weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) response (incidence and duration) | Baseline and 6-8 weeks post enrolment
  70% of patients (n = 36) had a >50% reduction in PSA from baseline.

SECONDARY OUTCOMES:
Radiologic response rate in patients with measurable disease | Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
  Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
PSA progression-free survival | Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
  Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
Disease progression-free survival | Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
  Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
Overall survival | Survival data collected to 100 weeks
  Median survival was 61 weeks and 1-year survival was 71%.
Safety and tolerability | Recruitment was stopped early due to elevated rates of febrile neutropenia. Safety data collected throughout duration.
  Recruitment was stopped due to higher than expected febrile neutropenia rate (27%). Fifty-one SAEs were reported in 33 patients, of which 7 were related to PI-88 treatment: non-neutropenic sepsis, neutropenic sepsis, pulmonary embolism, febrile dyspnoea, haematuria (x2), left middle cerebral artery infarction.
  Grade 3 or 4 AEs reported in >5% of patients comprise dehydration, fatigue, diarrhoea, nausea and thrombocytopenia.
  Two patients died during the study, one due to a ruptured abdominal aortic aneurysm, and one due to metastatic prostate cancer.
Quality of life Functional Assessment of Cancer Therapy - Prostate questionnaire (FACT-P) | Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
  Recruitment was stopped early due to elevated rates of febrile neutropenia. This end point was not reported.
Exploratory predictive value of biologic parameters C-reactive protein (CRP), vascular endothelial growth factor (VEGF), interleukin-6 (IL6), D-dimer | Baseline and 6-8 weeks post enrolment
  Change in VEGF trended towards prediction of survival (p = 0.056); pre-treatment and post-treatment levels of CRP were predictive of survival (p = 0.026, and p = 0.005 respectively) but the change in CRP was not (p = 0.999). IL-6 pretreatment levels were not predictive (p = 0.5111) but post-treatment (p = 0.0008) and change (p = 0.0020) were.
  These data need to interpreted with caution due to the small patient numbers involved.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Marx, MD, Study Chair — Sydney Haematology and Oncology Clinics; Nick Pavlakis, MD, Study Chair — Royal North Shore Hospital
Locations (8):
- Australia (8):
  - Sydney Haematology and Oncology Clinics, Hornsby, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Liverpool Cancer Therapy Centre, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Ashford Cancer Centre, Ashford, South Australia
  - Border Medical Oncology, Wodonga, Victoria

REFERENCES:
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213